CLINICAL TRIAL: NCT02657772
Title: Ultra Coils From Start to Finish for the Endovascular Repair of Small Intracranial Aneurysms
Acronym: ULTRA
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Stryker Neurovascular (Industry)
Responsible Party: Principal Investigator, Gaurav Jindal, Assistant Professor of Radiology, Neurosurgery, Neurology, University of Maryland, Baltimore
Other Study IDs: HP-00055046
Record Dates: First submitted 2016-01-14; First posted 2016-01-18 (Estimated); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Intracranial Aneurysms
Keywords: Target Ultra coils; small aneurysms
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess the safety and efficacy rates of the treatment of small intracranial aneurysms with Stryker Neurovascular's Target® 360 Ultra coils which are a type of platinum coils used to occlude aneurysms.

DETAILED DESCRIPTION:
This is a Prospective single-arm multi-center Registry which aims to collect data to determine the safety and efficacy of one of these marketed coils, namely the Target® 360 Ultra coils. This is not an intervention or treatment study. Up to 100 subjects at up to 6 sites will be enrolled.

Study Procedure

1. Screening and Informed consent: Patients will undergoing endovascular treatment of intracranial aneurysm will be screened using the Eligibility criteria checklist, and enrolled using approved Institutional Informed Consent process and approved Informed Consent form.
2. Baseline assessment: This involves standard of care history, medical examinations and laboratory assessments prior to coiling procedure.
3. Coiling procedure
4. One day post procedure assessment
5. 3- 28 days post procedure assessment
6. 3-9 months post procedure assessment
7. 9-18 months post procedure assessment

The Site investigator and/or co-investigator or their representative(s) will conduct training before initiating the study to develop a common understanding of the clinical protocol, Case Report Forms, and study procedures among the investigators and site research staff. Regulatory binders with study protocol, training documents, and standard operating guidelines will be provided for each study site. The Principal investigator and/or co-investigator shall confirm data received is accurate by reviewing with the provider collecting the data. The principle investigator and/or co-investigator will approve all data received. Additionally, OpenClinica, a web-based data capture service, will receive all Case Report Forms.

Study Monitoring will be electronic requiring upload of de-identified source documents through provided secure channels. However on site visits maybe scheduled in advance with the site personnel. Audits may be also be performed for quality assurance.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is between 18 and 80 years of age (inclusive).
2. Patient has a documented untreated intracranial aneurysm less than or equal to 5.0 mm in maximal dimension, ruptured or unruptured, suitable for embolization with coils.
3. Target® Ultra coils may be used.
4. Target aneurysm can be completely or nearly completely coiled at index procedure (No staged treatment procedures) without anticipated need for any target aneurysm reintervention after 72 hours of the index procedure. If a stent is to be placed during a separate preliminary procedure, then screening and enrollment for the coiling procedure must take place after the stenting procedure is completed.
5. Target aneurysm morphology allows for adequate retention of coils within the aneurysmal sac without occlusion of the parent artery, as determined by the treating physician.
6. Patient (or patient's legally authorized representative) has provided written informed consent.
7. Patient is willing and able to comply with protocol follow-up requirements.

Exclusion Criteria:

1. Patient is <18 or >80 years old.
2. Target aneurysm is felt by the physician operator to be mycotic or clearly dissecting in etiology.
3. Target aneurysm is >5.0 mm maximum luminal dimension.
4. Target aneurysm has been previously treated by surgery or endovascular therapy.
5. Target aneurysm is in the physician's estimation unlikely to be successfully treated by endovascular techniques.
6. Patient presents as Hunt and Hess grade V for a ruptured aneurysm.
7. Patient has known hypersensitivity to platinum, tungsten, nickel, stainless steel or structurally related compounds found in Target® Ultra coils.
8. Patients who have had or could have a severe reaction to contrast agents that cannot be adequately pre-medicated prior to the coiling procedure.
9. Patients who are unable to complete scheduled follow up assessments at the enrolling center due to limited life expectancy (<24 months), comorbidities or geographical considerations.
10. Patients with Moya-Moya disease, brain arteriovenous malformation(s), significant atherosclerotic stenosis, tortuousity or other conditions preventing access to the target aneurysm.
11. Target aneurysm with significant thrombosis that may increase the likelihood of recanalization at the discretion on the investigator.
12. Female patient has a positive pregnancy assessment at baseline, breastfeeding patient, or patient who plans to become pregnant within the 18 months following coiling.
13. The following comorbidities that may confound results: (a) organ failure of kidney (b) uncorrectable coagulation abnormality.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be between 18 and 80 years of age (inclusive)and have a documented untreated intracranial aneurysm, less than or equal to 5 mm, ruptured or unruptured, for which Ultra® coils are treatment options, and for which primary coiling treatment is planned to be completed during a single procedure (i.e., no "staged" treatment). Preliminary intracranial stent placement and/or use of an intracranial endoluminal balloon device as adjunctive therapy is allowed.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Target Aneurysm Recurrence (TAR) | 9-18 months from baseline/procedure date
  Target Aneurysm Recurrence (TAR) - defined as clinically relevant recurrence resulting in: target aneurysm re-intervention, rupture/re-rupture, and/or death from unknown cause as assessed at 9-18 months post procedure.

SECONDARY OUTCOMES:
Residual Aneurysm assessment using modified Raymond Scale | 9-18 months from baseline/procedure date
  Residual Aneurysm assessment using modified Raymond Scale (complete occlusion, minimal residual, residual aneurysm)
Modified Rankin Scale | Baseline, 1 Day post procedure, 3- 28 days post procedure, 3-9 months, 9-18 months from baseline/procedure date
  Assess the disability or degree of dependence of participants with Modified Rankin Scale score </=2 to determine good clinical outcomes at 9-18 months. It is compared with baseline values.
Technical procedural success | Procedure
  Technical procedural success defined as the successful delivery and deployment of Ultra® coils in the target aneurysm

CONTACTS AND LOCATIONS:
Overall Officials: Gaurav Jindal, MD, Principal Investigator — University of Maryland, Baltimore
Locations (6):
- United States (6):
  - Christiana Care Health System, Newark, Delaware
  - WellStar Research Institute, Marietta, Georgia
  - University of Maryland Baltimore, Baltimore, Maryland
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Geisinger medical center, Danville, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
The enrolled subjects will be assigned a unique research code that will not be associated with any identifiable information. All health information will be de-identified.

REFERENCES:
- [Derived] Jindal G, Almardawi R, Gupta R, Colby GP, Schirmer CM, Satti SR, Pukenas B, Hui FK, Caplan J, Miller T, Cherian J, Aldrich F, Kibria G, Simard JM; ULTRA Study Investigators. Target Ultra and Nano coils in the endovascular treatment of small intracranial aneurysms (ULTRA Registry). J Neurosurg. 2022 Jun 24;138(1):233-240. doi: 10.3171/2022.5.JNS2296. Print 2023 Jan 1. PMID 35901755